CLINICAL TRIAL: NCT06486974
Title: Efficacy of Manual Toothbrushes in Removing Tooth Stains: A 6-Week Clinical Research Study.
Brief Title: Efficacy of Manual Toothbrushes in Removing Tooth Stains
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-08-STN-DRW-DR-BGS
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Tooth Discoloration
Keywords: Lobene Tooth Stain Index
MeSH Terms: conditions — Tooth Discoloration | interventions — Supersmile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Colgate MaxFresh Toothpaste - 0.243% NaF (1100 ppm F)
  Total Polish 23 CHS TB Colgate Active Prevention Manual Toothbrush
  Interventions: Drug: NaF
- Group 2 (Active Comparator): Colgate Great Regular Flavor Toothpaste - 0.76% Na MFP (1000 ppm F)
  Colgate Adult Extra Clean soft-bristle toothbrush
  Interventions: Drug: Na MFP

INTERVENTIONS:
Drug: NaF — Group 1 will be instructed to brush their teeth twice daily/2 minutes each time for the duration of this study
  Arms: Group 1
Drug: Na MFP — Group 2 will be instructed to brush their teeth twice daily/2 minutes each time for the duration of this study
  Arms: Group 2

SUMMARY:
Efficacy of Manual Toothbrushes in Removing Tooth Stains: A 6-Week Clinical Research Study.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of manual toothbrushes in reducing tooth staining after 6 weeks of unsupervised, daily use by participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Male and female subjects, aged 18-70, inclusive;
* Good general health and good oral health based on the opinion of the study investigator;
* Presence of permanent natural anterior teeth (no veneers/crowns/restorations that may interfere with this study scoring procedures);
* A minimum composite mean of 1.5 ≥ determined by the Lobene Tooth Stain Index;
* Available for the duration of the study;
* Clinical evidence of a tendency to form extrinsic stains on anterior teeth.

Exclusion Criteria:

* Presence of orthodontic appliances/retainers involving scorable teeth;
* Presence of partial removable/fixed dentures and/or restorations involving scorable teeth;
* Tumor(s) of the soft or hard tissues of the oral cavity;
* Obvious signs of periodontal disease rampant caries, or any condition that the dental examiner considers exclusionary from the study;
* Five or more carious lesions requiring immediate care;
* Use of antibiotics, stain-inducing medications, and/or on any prescription that might interfere with the study outcome;
* Concurrent participation in another clinical study;
* Self-reported pregnancy and/or lactating women;
* Have used professional whitening product within one (1) year or had a dental prophylaxis (professional dental cleaning) within thirty (30) days - prior to the start of the study;
* History of allergies to oral care/personal care consumer products or their ingredients;
* History of alcohol and/or drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Lobene Tooth Stain Index | Baseline, and 6-weeks
  Each tooth will be scored separately using a 4 point area Stain Area (extent):
  (0) No stain detected
  1. Stain covering up to one third (1/3) of the region
  2. Stain covering > 1/3 to 2/3 of the region
  3. Stain covering > 2/3 of the region
  Stain Intensity:
  (0) No stain
  1. Light Stain - yellow to light brown or gray
  2. Moderate stain - medium brown
  3. Heavy stain - dark brown to black and intensity scale ranging from: Using the Lobene Tooth Stain Index, each tooth will be scored separately using a 4 point area and intensity scale ranging from:

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Garcia-Godoy, DDS, MS, PhD, Principal Investigator — Global Research Consultants
Locations (1):
- Spa Dental, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No